CLINICAL TRIAL: NCT03179852
Title: Effects of Nutrition Education on 3rd and 5th Grade Student's Fruit and Vegetable Consumption and Knowledge
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Washington University (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16124
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: nutrition education — nutrition education

SUMMARY:
The primary objective is to assess pre- and post-intervention nutrition education knowledge and preference. The secondary objective is to assess pre- and post-intervention fruit and vegetable consumption via a plate waste study.

DETAILED DESCRIPTION:
Background: The prevalence of overweight and obese children in the United States is at epidemic proportions, making it a recognized public health priority. Overweight and obese children are more likely to remain overweight and obese as adults, which increases their risk for developing obesity-related diseases and psychological disorders. Research shows that regular consumption of fruit and vegetables (F/V) may reduce the risk of obesity and obesity-related diseases yet most American school children fail to meet recommended intakes .

Objective: The purpose of this study was to determine if a F/V-targeted nutrition education intervention would increase F/V preference, knowledge, and consumption among elementary-school students.

Methods: Eight 20-minute nutrition lessons, focusing on F/V consumption, were administered over an eight-week period to 3rd and 5th grade students (N=150) at a local Ellensburg School District elementary school . Pre/post surveys were used to examine F/V knowledge and preference. Researchers observed and photographed students' lunches for 5-consecutive days pre- and post- intervention to assess possible change in consumption patterns.

Results: Data is currently under analysis. Conclusions: To be determined June 2017.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the National School Lunch Program

Exclusion Criteria:

* Did not participate in the National School Lunch Program

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in nutrition knowledge | Nutrition knowledge surveys will be administered during week 1 and again at week 10 after the 8 week nutrition education intervention
  surveys
Change in fruit and vegetable preferences | Fruit and vegetable preference surveys will be administered during week 1 and again at week 10 after the 8 week nutrition education intervention
  surveys

SECONDARY OUTCOMES:
Change in fruit and vegetable intake | Plate waste will be measured via the quarter waste method during week 1 and again at week 10 after the 8 week nutrition education intervention
  plate waste study

IPD SHARING:
Plan to Share IPD: No